CLINICAL TRIAL: NCT03999424
Title: The Safety and Efficacy of Autologous Human Schwann Cell (ahSC) Augmentation of Nerve Autografts After Severe Peripheral Nerve Injury (PNI)
Brief Title: Autologous Human Schwann Cells in Peripheral Nerve Repair
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: W. Dalton Dietrich (Other)
Collaborators: The Miami Project to Cure Paralysis (Other)
Responsible Party: Sponsor-Investigator, W. Dalton Dietrich, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20190453
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous human Schwann cells (Experimental): All participants will receive autologous human Schwann cells harvested from their own sural nerve.
  Interventions: Biological: autologous human Schwann cells

INTERVENTIONS:
Biological: autologous human Schwann cells — Schwann cells harvested from the sural nerve and debrided, injured sciatic nerve of the participant will be autologously transplanted along sural nerve autografts wrapped in a collagen matrix

SUMMARY:
The purpose of this study is to assess the safety of autologous human Schwann cell (ahSC) augmentation of nerve autograft repair in participants with severe peripheral nerve injury (PNI). For humans with acute severe PNI, the hypothesis is that augmentation of nerve autograft repair with ahSCs can potentially enhance axonal regeneration and myelin repair and thus improve functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Persons with severe sciatic nerve injury, brachial plexus injury, and/or major injury at the upper or lower extremity with nerve loss within previous year;
* Peripheral nerve injury with large gap (5 - 10 cm) between healthy nerve endings;
* Between the ages of 18 and 65 years at last birthday;

Exclusion Criteria:

* Persons unable to safely undergo an MRI (may include persons with an implanted device or metallic fragments which may interfere with MRI safety);
* Persons with pre-existing conditions that would preclude satisfactory sural nerve harvest (may include amputation or major injury to lower limb, or disease affecting the sural nerve);
* Persons with severe peripheral nerve injury gap length > 10 cm in length;
* Persons with history of radiation or local cancer in area of nerve injury, including primary tumors of the nerve;
* Pregnant women or a positive pregnancy test in those women with reproductive potential prior to transplantation;
* Presence of disease that might interfere with participant safety, compliance, or evaluation of the condition under study;
* History of active substance abuse;
* Persons allergic to gentamicin;
* Persons who test positive for HIV or Hepatitis B or C virus;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with reported adverse events (AEs) | 12 months post-transplantation
  The number of participants with reported AEs will be evaluated to assess safety. Using CTCAE v4.0 grading scale, all AEs that are Grade 3 or higher with treating physician's attribution of probable or definite relation to intervention will be included.
Number of participants with reported cell product culture test failure | 12 months post-transplantation
  Using sterility testing, the number of participants with reported cell product culture test failure will be evaluated.
Change in muscle strength scale grade of affected limb muscles | from baseline to 12 months post-transplantation
  The Medical Research Council (MRC) scale for muscle strength grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Sensory recovery scale grade of affected dermatomes | from baseline to 12 months post-transplantation
  Assessment of pin-prick and two point discrimination in areas previously anesthetic in the distal distribution of the nerve injury.
Change in pain scores | from baseline to 12 months post-transplantation
  The Douleur Neuropathique 4 (DN4) questionnaire estimates the probability of neuropathic pain, based on 10 items. Seven items related to pain quality are based on an interview and 3 items are based on clinical examination.
Change in pain characteristics (location, intensity, and description) | from baseline to 12 months post-transplantation
  Assessed by a pain diagram which identifies areas of pain with descriptors. An intensity scale from 0 (no pain) to 10 (most intense pain imaginable) is used to rate the overall intensity of pain at the time of assessment.
Number of participants with reported tumorigenesis or unexpected changes in nerve structure | 2 years post-transplantation
  Tumorigenesis and/or unexpected changes in the nerve structure will be determined by evaluation of magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Change in muscle strength scale grade of affected limb muscles | from baseline to 5 years
  The Medical Research Council (MRC) scale for muscle strength grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Sensory recovery scale grade of affected dermatomes | from baseline to 5 years
  Assessment of pin-prick and two point discrimination in areas previously anesthetic in the distal distribution of the nerve injury.
Change in pain scores | from baseline to 5 years post-transplantation
  The Douleur Neuropathique 4 (DN4) questionnaire estimates the probability of neuropathic pain, based on 10 items. Seven items related to pain quality are based on an interview and 3 items are based on clinical examination.
Change in pain characteristics (location, intensity, and description) | from baseline to 5 months post-transplantation
  Assessed by a pain diagram which identifies areas of pain with descriptors. An intensity scale from 0 (no pain) to 10 (most intense pain imaginable) is used to rate the overall intensity of pain at the time of assessment.
Nerve-graft continuity | 2 weeks post-transplantation
  Ultrasound will be used to assess nerve-graft continuity.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Levi, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No